CLINICAL TRIAL: NCT01502488
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intravenously in Patients With Autism
Brief Title: Adipose Derived Stem Cell Therapy for Autism
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-AT-001
Record Dates: First submitted 2011-12-27; First posted 2011-12-30 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Autism
Keywords: Autistic; ASC therapy; ADSC
MeSH Terms: conditions — Autistic Disorder | interventions — Lipectomy; HMGA2 Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Fat Harvesting and Stem Cell Injection — Cells will be harvested through a local liposuction and injected via IV delivery
  Other Names: Liposuction; Adipose Derived Stem Cell Injection; ADSC; Lipo; Fat Stem Cells; IV

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients with Autism.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of ASC implantation after liposuction using an IV delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 and 12 years.
* DSM-IV diagnosis of Autistic Disorder.
* Total score of CARS ≥ 30.
* Parents or legal guardian willing to sign the ICF.

Exclusion Criteria:

* History of prior or current DSM-IV psychotic disorder (e.g., schizophrenia, bipolar disorder, other psychosis), Pervasive Developmental Disorder not otherwise specified (PDD NOS), Asperger's, or Rett's.
* History of Epileptic seizure activity in the past 6 months.
* Autism caused by seizure disorders (active), cerebrovascular disease or brain trauma.
* The global autism ratings are assessed as being absent, minimal or mild.
* Existing moderate or severe extrapyramidal symptoms (EPS) or history of tardive dyskinesia.
* Active infectious disease and/or known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will have expert consultation to determine eligibility based on the patient's infectious status
* Enrollment in other trials in the last 3 months without agreement to discontinue them.
* Life expectancy < 6 months due to concomitant illnesses.
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Active clinical infection within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer
* Parental unwillingness and/or not able to give written informed consent.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in the Childhood Autism Rating Scale，CARS | 3 months
Improvement in the Clinical Global Impression Scale, CGI | 3 months
Improvement in the Childhood Autism Rating Scale，CARS | 6 months
Improvement in the Clinical Global Impression Scale, CGI | 6 months

SECONDARY OUTCOMES:
Improvement in the Aberrant Behavior Checklist, ABC | 3 months
Improvement in the Aberrant Behavior Checklist, ABC | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided